CLINICAL TRIAL: NCT05282173
Title: Training CHWs to Support Re-Engagement in TB/HIV Care in the Context of Depression and Substance Use
Brief Title: Community Health Worker Training to Reduce Depression and Substance Use Stigma in TB/HIV Care in South Africa
Acronym: Siyakhana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Medical Research Council, South Africa (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: EC039-10/2021; R34MH122268 (NIH)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Substance-Related Disorders; Mental Disorder; Social Stigma; Depression; Treatment Adherence and Compliance; Health Care Utilization; Attitude of Health Personnel; Hiv; Tuberculosis; Mental Health Disorder; Community Health Workers; Health Care Delivery
Keywords: Substance-Related Disorders; Mental Disorders; Social Stigma; Depression; Treatment Adherence and Compliance; Delivery of Health Care; Attitude of Health Personnel; HIV; Tuberculosis; Health Care Utilization; Mental Health; Global Health; South Africa; Community Health Workers
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders; Social Stigma; Depression; Treatment Adherence and Compliance; Patient Acceptance of Health Care; Acquired Immunodeficiency Syndrome; Tuberculosis; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study uses a stepped-wedge design. All groups of CHWs receive both treatment as usual (TAU) and the stigma reduction training ("Siyakhana"). Randomization will dictate the timing/order in which each group receives the Siyakhana training.
Masking Description: The staff member who conducts role-play assessments with participants will be minimally involved in the Siyakhana training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): Monitoring of treatment as usual (i.e., routine interactions between community health workers (CHWs) and their patients).
- Siyakhana CHW Training (Experimental): The Siyakhana CHW Training is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
  Interventions: Behavioral: Siyakhana CHW Training

INTERVENTIONS:
Behavioral: Siyakhana CHW Training — Please see arm description.
  Other Names: Siyakhana; Siyakhana - C
  Arms: Siyakhana CHW Training

SUMMARY:
Poor engagement in care contributes to HIV- and TB-related morbidity and mortality in South Africa (SA). Community health workers (CHWs) are frontline lay health workers who work to re-engage patients who are lost to follow-up (LTFU) in HIV/TB care. Patients with depression and substance use (SU) have a greater likelihood of being LTFU in HIV/TB care, and there is evidence that CHWs may exhibit stigma towards these patients. When CHWs have negative attitudes towards these patients, on average they spend less time with these patients, are less likely to implement evidence-based practices, and deliver less patient-centered care. Therefore, this purpose of this study is to examine the implementation and preliminary effectiveness of a brief training ("Siyakhana"). The purpose of this training is to provide CHWs with psychoeducation, skills, and support around working with HIV/TB patients with depression/SU. The investigators will assess the training's implementation and changes in CHWs' stigma towards HIV/TB patients with depression/SU.

DETAILED DESCRIPTION:
South Africa (SA) has the highest number of people living with HIV in the world and a high tuberculosis (TB) burden. Poor engagement in care contributes to HIV- and TB-related morbidity and mortality. In this context, community health workers (CHWs) are frontline lay health workers who play a central role in re-engaging patients who are lost to follow-up (LTFU) in HIV/TB care. Even with existing CHW programs focused on re-engaging patients who are LTFU, people with depression, hazardous alcohol use, or other substance use (SU) are particularly susceptible to poor engagement in HIV/TB care and have a greater likelihood of being LTFU. At the moment, CHWs receive minimal, if any, training on depression and SU, and there is some evidence that CHWs may exhibit stigma towards these patients. When CHWs have negative attitudes towards these patients, on average they spend less time with these patients, are less likely to implement evidence-based practices, and deliver less patient-centered care. Therefore, the purpose of this study is to examine the implementation and preliminary effectiveness of a brief training ("Siyakhana") focused on providing CHWs with psychoeducation, skills, and support around working with patients with depression/SU. In a Type 2, hybrid effectiveness-implementation trial, and using a stepped wedge design, the investigators will primarily assess the training's implementation (feasibility, acceptability, and fidelity) and changes in CHWs' stigma towards HIV/TB patients with depression/SU.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Employed as a CHW through a partner non-governmental organization (NGO) that provides HIV/TB CHW services
* Works with patients who have HIV and TB, some of whom may be struggling with depression or substance use

Exclusion Criteria:

* Unable to complete informed consent or study procedures in English or Xhosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, PhD, Principal Investigator — University of Maryland; Bronwyn J Myers, PhD, Principal Investigator — Medical Research Council, South Africa
Locations (1):
- South African Medical Research Council, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be available per request of outside individual.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study has been complete (all data collected; data analysis only), the Study Protocol, Informed Consent Forms (ICFs), and Statistical Analysis Plan (SAP) will be made available per request of outside individual.
Access Criteria: Supporting information will be made available per request of outside individuals.

REFERENCES:
- [Derived] Magidson JF, Regenauer KS, Johnson K, Ma T, Belus JM, Rose AL, Brown I, Ciya N, Ndamase S, Sacko C, Joska J, Sibeko G, Bassett IV, Myers B. Siyakhana: A hybrid type 2 effectiveness-implementation stepped-wedge trial to reduce stigma towards substance use and depression among community health workers in HIV/TB care in South Africa. J Subst Use Addict Treat. 2025 Apr;171:209634. doi: 10.1016/j.josat.2025.209634. Epub 2025 Jan 31. PMID 39892671
- [Derived] Myers B, Regenauer KS, Rose A, Johnson K, Ndamase S, Ciya N, Brown I, Joska J, Bassett IV, Belus JM, Ma TC, Sibeko G, Magidson JF. Community health worker training to reduce mental health and substance use stigma towards patients who have disengaged from HIV/TB care in South Africa: protocol for a stepped wedge hybrid type II pilot implementation trial. Implement Sci Commun. 2024 Jan 2;5(1):1. doi: 10.1186/s43058-023-00537-w. PMID 38167261

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Sequence 1: Approximately 1 Month Treatment as Usual, Siyakhana CHW Training: Group 1 was randomized to receive approximately 1-month of TAU then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
- Sequence 2: Approximately 2 Months Treatment as Usual, Siyakhana CHW Training: Group 2 was randomized to receive approximately two-months of treatment as usual (TAU) then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
  Siyakhana CHW Training: Please see arm description.
- Sequence 3: Approximately 3 Months Treatment as Usual, Siyakhana CHW Training: Group 3 was randomized to receive approximately 3-months of TAU then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
Period: Overall Study
Arm/Group | Sequence 1: Approximately 1 Month Treatment as Usual, Siyakhana CHW Training | Sequence 2: Approximately 2 Months Treatment as Usual, Siyakhana CHW Training | Sequence 3: Approximately 3 Months Treatment as Usual, Siyakhana CHW Training
Started | 29; 2 Clinics | 25; 2 Clinics | 28; 2 Clinics
Completed | 26; 2 Clinics | 23; 2 Clinics | 24; 2 Clinics
Not Completed | 3; 0 Clinics | 2; 0 Clinics | 4; 0 Clinics
Not completed — Missed | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Arm/Group | Siyakhana CHW Training
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 82
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 82
CHW Substance Use Stigma [Mean (Standard Deviation); unit: units on a scale] — CHW stigma towards substance use was measured using the Social Distance Scale (SDS). SDS scores range from 6 to 24, with higher scores indicating more desired social distance (more stigma).
  units on a scale | 12.53 (3.44)
CHW Depression Stigma [Mean (Standard Deviation); unit: units on a scale] — CHW stigma towards depression was measured using the Social Distance Scale (SDS). SDS scores range from 6 to 24, with higher scores indicating more desired social distance (more stigma).
  units on a scale | 8.33 (2.17)

OUTCOME MEASURES:

1. Primary Outcome: CHW Stigma Towards Substance Use
Description: CHW stigma towards substance use measured using the Social Distance Scale (SDS). SDS scores range from 6 to 24, with higher scores indicating more desired social distance (more stigma).
Time Frame: Change between baseline assessment and 6-month follow-up (approximately 6-months post-training)
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | Siyakhana CHW Training
Number analyzed (Participants) | 73
change in units on a scale | -0.88 (0.39)

2. Primary Outcome: CHW Stigma Towards Depression
Description: CHW stigma towards depression measured using the Social Distance Scale (SDS). SDS scores range from 6 to 24, with higher scores indicating more desired social distance (more stigma).
Time Frame: Change between baseline assessment and 6-month follow-up (approximately 6-months post-training)
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | Siyakhana CHW Training
Number analyzed (Participants) | 73
change in units on a scale | 0.15 (0.73)

3. Primary Outcome: Training Feasibility
Description: The number of CHWs who attended all three days of the Siyakhana training. The training will be considered feasible if over 75% of CHWs attend the full training.
Time Frame: 3-months post-training
Measure: Count of Participants; unit: Participants
Groups:
- Sequence 2: Approximately 2 Months TAU, Siyakhana CHW Training: Group 2 was randomized to receive approximately 2-months of TAU then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
- Sequence 3: Approximately 3 Months TAU, Siyakhana CHW Training: Group 3 was randomized to receive approximately 3-months of TAU then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
Arm/Group | Sequence 1: Approximately 1 Month Treatment as Usual, Siyakhana CHW Training | Sequence 2: Approximately 2 Months TAU, Siyakhana CHW Training | Sequence 3: Approximately 3 Months TAU, Siyakhana CHW Training
Number analyzed (Participants) | 29 | 25 | 28
Participants | 26 | 25 | 27

4. Primary Outcome: Acceptability
Description: Acceptability subscale of the John Hopkins D&I Measure, a 12-item measure for assessing dissemination and implementation outcomes in low- and middle-income settings. This measure will specifically assess CHW's perceived satisfaction, relevance, usefulness, comprehension, and comfort level of the training. Items are rated on a 0-3 scale, and averaged, with lower scores (closer to 0) indicating low acceptability and higher scores (closer to 3) indicating higher acceptability.
Time Frame: 3-months post-training
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sequence 1: Approximately 1 Month TAU, Siyakhana CHW Training: Group 1 was randomized to receive approximately 1-month of TAU then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
- Sequence 3: Approximately 3 Months TAU, Siyakhana CHW Training: Group 13 was randomized to receive approximately 3-months of TAU then the Siyakhana CHW Training, which is a multi-day group training that aims to reduce stigma around mental health and substance use among CHWs. It integrates psychoeducation around TB/HIV, stigma, depression, and substance use, including countering myths and stereotypes around mental health and substance use; skills for CHW self-care; evidence-based skills for working with patients living with depression and substance use, such as components of motivational interviewing and problem-solving therapy; and exposure to individuals with lived experience of mental health and substance use. The training is a combination of informative presentations, discussions, worksheets/activities, and role-plays aimed at increasing awareness of mental health and substance use, reducing stigma, and improving interactions when working with patients with HIV/TB and mental health and substance use concerns.
Arm/Group | Sequence 1: Approximately 1 Month TAU, Siyakhana CHW Training | Sequence 2: Approximately 2 Months TAU, Siyakhana CHW Training | Sequence 3: Approximately 3 Months TAU, Siyakhana CHW Training
Number analyzed (Participants) | 27 | 23 | 25
units on a scale | 2.92 (0.29) | 2.84 (0.26) | 2.80 (0.24)

5. Primary Outcome: CHW Training Fidelity
Description: 20% of CHW role-plays at the 3-month follow-up assessment (approximately 3-months post-training) randomly selected for rating using the ENhancing Assessment of Common Therapeutic factors (ENACT) tool, a 15-item validated measure of fidelity and clinical competence among non-specialist workers, by two independent bilingual assessors. Ratings were given for 15 clinical competencies, giving scores of 1 (harmful), 2 (some basic skills), 3 (all basic skills), or 4 (advanced skills). CHW fidelity scores were calculated based on ENACT items rated as delivered with competence. A cut-off of ≥2 (some basic skills) was used to define fidelity for each item.
Time Frame: 3-months post-training
Population: Note the fidelity measure is a randomly selected 20% of roleplays that were coded by an independent rater across all sessions.
Measure: Mean (Standard Deviation); unit: % of components delivered competently
Arm/Group | Sequence 1: Approximately 1 Month TAU, Siyakhana CHW Training | Sequence 2: Approximately 2 Months TAU, Siyakhana CHW Training | Sequence 3: Approximately 3 Months TAU, Siyakhana CHW Training
Number analyzed (Participants) | 29 | 25 | 28
% of components delivered competently | 86.7 (8.2) | 85.7 (11.8) | 82.7 (10.1)

6. Secondary Outcome: CHW Stigma Towards Substance Use
Description: as for outcome 1
Time Frame: Change between baseline assessment and 3-month follow-up (approximately 3-months post-training)
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | Siyakhana CHW Training
Number analyzed (Participants) | 77
change in units on a scale | -1.22 (0.35)

7. Secondary Outcome: CHW Stigma Towards Depression
Description: as for outcome 2
Time Frame: Change between baseline assessment and 3-month follow-up (approximately 3-months post-training)
Measure: Mean (Standard Error); unit: change in units on a scale
Arm/Group | Siyakhana CHW Training
Number analyzed (Participants) | 77
change in units on a scale | 0.51 (1.17)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition for AE and/or SAE did not differ from the clinicaltrials.gov definition.
Arm/Group | Sequence 1: Approximately 1 Month TAU, Siyakhana CHW Training | Sequence 2: Approximately 2 Months TAU, Siyakhana CHW Training | Sequence 3: Approximately 3 Months TAU, Siyakhana CHW Training
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT05282173/Prot_SAP_000.pdf